CLINICAL TRIAL: NCT00111085
Title: A Phase IIb, Multi-center, International, Double-blind, Randomized, Placebo-controlled, Parallel-group, Dose-finding Study for the Prevention of Cerebral Vasospasm After Aneurysmal Subarachnoid Hemorrhage (aSAH) by Intravenous Administration of Clazosentan, a Selective Endothelin A (ETA) Receptor Antagonist
Brief Title: Clazosentan in Preventing the Occurrence of Cerebral Vasospasm Following an Aneurysmal Subarachnoid Hemorrhage (aSAH)
Acronym: CONSCIOUS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: AC-054-201
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: delayed ischemic neurological deficits (DIND); vasospasm; clazosentan; cerebral vasospasm; computer tomography scan (CT scan); digital subtraction angiography (DSA); endothelin A receptor; aneurysmal subarachnoid hemorrhage (aSAH)
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — clazosentan

ARMS (4):
- Clazosentan 1 mg/h (Experimental): intravenous clazosentan at 1 mg/h starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Interventions: Drug: Clazosentan 1 mg/h
- Clazosentan 5 mg/h (Experimental): intravenous clazosentan at 5 mg/h starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Interventions: Drug: Clazosentan 5 mg/h
- Clazosentan 15 mg/h (Experimental): intravenous clazosentan at of 15 mg/h starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Interventions: Drug: Clazosentan 15 mg/h
- Placebo (Placebo Comparator): intravenous placebo starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clazosentan 1 mg/h — Subjects receive intravenous clazosentan at a rate of 1 mg/h starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Other Names: ACT-108475
  Arms: Clazosentan 1 mg/h
Drug: Clazosentan 5 mg/h — Subjects receive intravenous clazosentan at a rate of 5 mg/h starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Other Names: ACT-108475
  Arms: Clazosentan 5 mg/h
Drug: Clazosentan 15 mg/h — Subjects receive intravenous clazosentan at a rate of 15 mg/h starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Other Names: ACT-108475
  Arms: Clazosentan 15 mg/h
Drug: Placebo — Subjects receive intravenous placebo starting within 56 hours maximum after aneurysm rupture and continuing until Day 14 post-aneurysm rupture
  Arms: Placebo

SUMMARY:
The purpose of the study is to measure how effective and safe three different doses of the drug clazosentan are in preventing vasospasm after subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged 18 to 70 years (inclusive) or male patients aged 45 to 70 (inclusive) or males aged 18 to 44 (inclusive) who are surgically or naturally sterile or can personally sign the core Informed Consent
2. Patients with a ruptured saccular aneurysm that has been confirmed by digital subtraction angiography (DSA) and for which clipping or coiling (endovascular obliteration) is possible.
3. Patients with a diffuse or localized thick subarachnoid clot on baseline CT scan. Measurements defining clot thickness and extension are as follows: Diffuse: Clot with long axis >= 20 mm, or any clot if present in both hemispheres Localized: Clot with long axis < 20 mm Thick: Clot with short axis >= 4 mm Thin: Clot with short axis < 4 mm
4. Start of screening within 48 hours post onset of aSAH clinical symptoms
5. World Federation of Neurological Surgeons (WFNS) Grades I-IV, and those Grade V patients who improve to Grade IV or less after ventriculostomy
6. In the case of multiple aneurysms, the aneurysm that has ruptured is identified with a high likelihood during the screening period
7. Women of childbearing potential with pre-treatment negative serum pregnancy test
8. Patient is able to start the study drug infusion within 56 hours after the rupture of the aneurysm, and the procedure option (clipping or coiling) must either be started within a maximum of 12 hours after the start of study drug infusion or should have been already performed
9. Written informed consent to participate in the study must be obtained from the patient or a legal representative prior to initiation of any study-related procedure and enrollment

Exclusion criteria:

1. Patients with SAH due to other causes (e.g., trauma or rupture of fusiform or mycotic aneurysms)
2. Patients with intraventricular or intracerebral blood, in the absence of subarachnoid blood
3. No visualized clot or presence of only localized thin clot on CT (< 20 mm x 4 mm)
4. Presence of any degree of cerebral vasospasm on screening angiogram
5. Patients with hypotension (systolic blood pressure (SBP) <=90 mmHg) refractory to fluid therapy
6. Patients with neurogenic pulmonary edema or severe cardiac failure requiring inotropic support
7. Any severe or unstable concomitant condition or disease (e.g., known significant neurological deficit, cancer, hematological, or coronary disease), or chronic condition (e.g., psychiatric disorder) which, in the opinion of the Investigator, would affect the assessment of the safety or efficacy of the study drug
8. Advanced kidney and/or liver disease, as defined by plasma creatinine >=2 mg/dl (177 micromol/l) and/or total bilirubin > 3 mg/dl (51.3 micromol/l)
9. Any known or CT evidence of previous major cerebral damage (e.g., stroke [> 2 cm], traumatic brain injury [> 2 cm], previously treated cerebral aneurysm, arterial venous malformation [AVM]), or other preexisting cerebrovascular disorders, which may affect accurate diagnosis and evaluation of SAH
10. Patients receiving prophylactic i.v. nimodipine or i.v. nicardipine. If present, these must be stopped at least 4 hours prior to initiation of the study treatment
11. Patients who have received thrombolytics, including intracisternal administration, intrathecal treatments and therapeutic hypothermia for treatment of the SAH
12. Patients who have received an investigational product within 28 days prior to randomization
13. Patients with current alcohol or drug abuse or dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2005-01-10 (Actual); Primary Completion 2006-03-30 (Actual); Study Completion 2006-03-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of moderate or severe cerebral vasospasm, as measured by cerebral angiography | Up to day 14
  If the patient develops clinical or sonographic changes suggestive of vasospasm prior to or after Day 9 ± 2 and until Day 14 post-aneurysm rupture, an angiogram will be performed to confirm the vasospasm. If vasospasm is documented prior to Day 9 ± 2, the Day 9 ± 2 angiogram is no longer required. In the case that a patient only develops clinical symptoms suggestive of vasospasm later than Day 9 ± 2 and up to Day 14, an additional angiogram should be performed to confirm the diagnosis of vasospasm. If the latter shows a higher grade of vasospasm than the previous one, it will be used for comparison to the baseline angiogram for evaluation of the primary endpoint.

SECONDARY OUTCOMES:
Occurrence of vasospasm-related morbidity, and mortality of all causes defined as the occurrence of death of any cause within the first 6 weeks post-aneurysm rupture OR | Within 6 weeks
Occurrence of vasospasm-related morbidity, and mortality of all causes defined as the occurence of new cerebral infarct within first 6 weeks post-aneurysm rupture based on local investigator reading of post-baseline CT scans OR | Within 6 weeks
Occurrence of vasospasm-related morbidity, and mortality of all causes defined as the occurence of delayed ischemic neurological deficits (DIND) due to vasospasm (based on investigator assessments) within 14 days post-aneurysm rupture OR | Within 14 days
Occurrence of vasospasm-related morbidity, and mortality of all causes defined as occurrence of use of rescue medication due to vasospasm within 14 days post-aneurysm rupture | Within 14 days
Clinical outcome at 12 weeks post-aneurysm rupture as measured by the Modified Rankin Scale (mRS) score | At 12 weeks
Clinical outcome at 12 weeks post-aneurysm rupture as measured bythe Glasgow Outcome Scale - Extended Version (GOSE) score | At 12 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (10):
  - Dr. Giuseppe Lanzino, Peoria, Illinois
  - Dr. Horner, Indianapolis, Indiana
  - Dr. Aldrich, Baltimore, Maryland
  - Dr. Ogilvy, Boston, Massachusetts
  - Dr. Zuccarello, Cincinnati, Ohio
  - Dr. Woo, Cleveland, Ohio
  - Dr. Rosenwasser, Philadelphia, Pennsylvania
  - Dr. Zager, Philadelphia, Pennsylvania
  - Dr. George A. Lopez, Houston, Texas
  - Dr. Bullock, Richmond, Virginia
- Canada (6):
  - Dr. Wong, Calgary, Alberta
  - Dr. Findlay, Edmonton, Alberta
  - Dr. Redekop, Vancouver, British Columbia
  - Dr. Ferguson, Toronto, Ontario
  - Dr. Bojanowski, Montreal, Quebec
  - Dr. Fleetwood, Halifax, Nova Scotia

REFERENCES:
- [Derived] Eagles ME, Powell MF, Ayling OGS, Tso MK, Macdonald RL. Acute kidney injury after aneurysmal subarachnoid hemorrhage and its effect on patient outcome: an exploratory analysis. J Neurosurg. 2019 Jul 12;133(3):765-772. doi: 10.3171/2019.4.JNS19103. Print 2020 Sep 1. PMID 31299650
- [Derived] Ayling OGS, Ibrahim GM, Alotaibi NM, Gooderham PA, Macdonald RL. Anemia After Aneurysmal Subarachnoid Hemorrhage Is Associated With Poor Outcome and Death. Stroke. 2018 Aug;49(8):1859-1865. doi: 10.1161/STROKEAHA.117.020260. PMID 29946013
- [Derived] Ayling OG, Ibrahim GM, Alotaibi NM, Gooderham PA, Macdonald RL. Dissociation of Early and Delayed Cerebral Infarction After Aneurysmal Subarachnoid Hemorrhage. Stroke. 2016 Dec;47(12):2945-2951. doi: 10.1161/STROKEAHA.116.014794. Epub 2016 Nov 8. PMID 27827324
- [Derived] Nassiri F, Ibrahim GM, Badhiwala JH, Witiw CD, Mansouri A, Alotaibi NM, Macdonald RL. A Propensity Score-Matched Study of the Use of Non-steroidal Anti-inflammatory Agents Following Aneurysmal Subarachnoid Hemorrhage. Neurocrit Care. 2016 Dec;25(3):351-358. doi: 10.1007/s12028-016-0266-6. PMID 27000643
- [Derived] Tso MK, Ibrahim GM, Macdonald RL. Predictors of Shunt-Dependent Hydrocephalus Following Aneurysmal Subarachnoid Hemorrhage. World Neurosurg. 2016 Feb;86:226-32. doi: 10.1016/j.wneu.2015.09.056. Epub 2015 Sep 30. PMID 26428322
- [Derived] Young JM, Morgan BR, Misic B, Schweizer TA, Ibrahim GM, Macdonald RL. A Partial Least-Squares Analysis of Health-Related Quality-of-Life Outcomes After Aneurysmal Subarachnoid Hemorrhage. Neurosurgery. 2015 Dec;77(6):908-15; discussion 915. doi: 10.1227/NEU.0000000000000928. PMID 26248048
- [Derived] Ibrahim GM, Macdonald RL. The network topology of aneurysmal subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2015 Aug;86(8):895-901. doi: 10.1136/jnnp-2014-308992. Epub 2014 Oct 3. PMID 25280913
- [Derived] Ibrahim GM, Morgan BR, Macdonald RL. Patient phenotypes associated with outcomes after aneurysmal subarachnoid hemorrhage: a principal component analysis. Stroke. 2014 Mar;45(3):670-6. doi: 10.1161/STROKEAHA.113.003078. Epub 2014 Jan 14. PMID 24425125
- [Derived] Ibrahim GM, Fallah A, Macdonald RL. Clinical, laboratory, and radiographic predictors of the occurrence of seizures following aneurysmal subarachnoid hemorrhage. J Neurosurg. 2013 Aug;119(2):347-52. doi: 10.3171/2013.3.JNS122097. Epub 2013 Apr 12. PMID 23581590
- [Derived] Ibrahim GM, Macdonald RL. Electrocardiographic changes predict angiographic vasospasm after aneurysmal subarachnoid hemorrhage. Stroke. 2012 Aug;43(8):2102-7. doi: 10.1161/STROKEAHA.112.658153. Epub 2012 Jun 7. PMID 22678087
- [Derived] Ibrahim GM, Weidauer S, Vatter H, Raabe A, Macdonald RL. Attributing hypodensities on CT to angiographic vasospasm is not sensitive and unreliable. Stroke. 2012 Jan;43(1):109-12. doi: 10.1161/STROKEAHA.111.632745. Epub 2011 Oct 13. PMID 21998061